CLINICAL TRIAL: NCT00923026
Title: Follow-Up Protocol for Subjects Previously Enrolled on NCI Surgery Branch Studies
Brief Title: Follow Up Protocol for Subjects Previously Enrolled on NCI Surgery Branch Studies
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090161; 09-C-0161
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01-22

CONDITIONS: Melanoma; Adenocarcinoma; Carcinoma NOS; Neuroendocrine Tumors
Keywords: Gene Therapy; Follow-Up; Delayed Toxicity; Natural History; Adenocarcinoma; Melanoma; Neuroendocrine Tumors; Carcinoma
MeSH Terms: conditions — Melanoma; Adenocarcinoma; Carcinoma; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A/Gene Therapy: Patients who have received gene therapy
- B/Non-Gene Therapy: Patients who have not received gene therapy

SUMMARY:
Background:

The NCI Surgery Branch has developed experimental therapies that involve taking white blood cells from participants' tumor or from their blood, growing them in the laboratory in large numbers, and then giving the cells back to the patient.

Objective:

This study will allow participants to be followed for up to 15 years following treatment on an NCI Surgery Branch Gene Therapy Trial as required by the FDA.

Eligibility:

Participants must have been enrolled on an NCI Surgery Branch Gene Therapy Protocol

Design

Participants will be followed with a physical examination and blood tests for up to 15 years as required by the FDA

...

DETAILED DESCRIPTION:
Background:

* Patients receiving care at the NIH Clinical Center are required to be enrolled on a clinical protocol.
* Following participation in a treatment protocol, it may be in the best interest of the patient to continue to be followed at the Clinical Center.
* The National Cancer Institute Surgery Branch (NCI-SB) conducts clinical trials utilizing gene transfer. The current U.S. Food and Drug Administration (FDA) requirements for long-term follow-up are up to fifteen years for some products. As this time-period is frequently longer than studies are expected to be open, a long-term follow-up protocol is necessary to ensure the follow-up of these participants.

Objective:

-Primary objective:

--Provide a mechanism for long-term follow-up of participants who have participated in research studies in the NCI-SB.

Eligibility:

* Age greater than or equal to 18 years.
* Participant has been enrolled on an NCI-SB treatment protocol.

Design:

* Participant will undergo physical exams, laboratory evaluation, imaging, or phone follow-up as clinically indicated.
* Procedures that entail more than minimal risk to the patient should not be performed for research purposes on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years.
* Participants who have received treatment on an NCI-SB protocol, including gene therapy protocols. (Note: Participants may be enrolled on this protocol and, at the same time, participate in an active treatment study).
* For Cohort A:Ability of participant or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document. For Cohort B: Participant is able to provide informed consent.

EXCLUSION CRITERIA:

-For Cohort B: Individuals of child-bearing potential (IOCBP) who are pregnant or plan to become pregnant because of the potentially dangerous effects of the investigational treatments administered on NCI-SB treatment protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects will have previously been enrolled on an NCI Surgery Branch treatment protocol. Patients who received gene therapy will be followed as required by the FDA.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2009-06-15 (Actual)

PRIMARY OUTCOMES:
Long-term follow-up | Until time of death
  Long-term follow-up of subjects who have participated in research studies in the NCI Surgery Branch

SECONDARY OUTCOMES:
Long-term follow-up for gene therapy studies | 15 years
  Collection of long-term, follow-up information on subjects who have participated in gene transfer studies as required by the FDA and other regulatory groups
Survival | Until time of death
  Follow subjects who have participated in research studies in the NCI Surgery Branch until time of death

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-C-0161.html